CLINICAL TRIAL: NCT01421199
Title: A Prospective, Multi Center, Non-randomized Clinical Trial to Evaluate the Ear Effusion Detection and Characterization System (EEDCS) to Detect and Characterize Middle Ear Fluid in Children
Brief Title: Device Study to Evaluate the Detection and Characterization of Middle Ear Fluid in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: OtoSonics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: OTO-Myr
Record Dates: First submitted 2011-08-18; First posted 2011-08-22 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-08

CONDITIONS: Otitis Media With Effusion; Middle Ear Effusion
Keywords: Otitis Media with Effusion; Middle Ear Effusion
MeSH Terms: conditions — Otitis Media with Effusion | interventions — Middle Ear Ventilation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myringotomy (Other): On arm
  Interventions: Procedure: Myringotomy

INTERVENTIONS:
Procedure: Myringotomy — tube placement for children with multiple ear infections
  Other Names: ear tubes

SUMMARY:
The study has three objectives:

1. To determine if the device can detect if middle ear fluid is present in children who are scheduled for tube placement (myringotomy)
2. If fluid is present to characterize the fluid as thick or thin
3. Evaluate the safety of the device

ELIGIBILITY:
Inclusion Criteria:

* 6 months to 17 years
* scheduled to undergo myringotomy procedure

Exclusion Criteria:

* mastoiditis
* tympanostomy tubes
* chronic middle ear disease
* otitis externa
* perforations of the middle ear
* use of antibiotic ear drops within 2 days of surgery
* systemic antibiotic use

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 125 (Estimated)
Dates: Start 2011-09; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
detection of middle ear fluid | day one
  device will be used during myringotomy procedure to detect middle ear fluid

SECONDARY OUTCOMES:
fluid viscosity | day one
  fluid obtained during myringotomy will be tested for viscosity

CONTACTS AND LOCATIONS:
Overall Officials: Mark E Boseley, MD, Principal Investigator — Madigan Army Medical Center